CLINICAL TRIAL: NCT03155022
Title: Combined Application of Remote and Intra-Coronary Ischemic Conditioning in Acute Myocardial Infarction: A Multicenter, Randomized, Controlled Clinical Trial (CARIOCA Study)
Brief Title: Combined Application of Remote and Intra-Coronary Ischemic Conditioning in Acute Myocardial Infarction
Acronym: CARIOCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL17_0032; 2017-A01683-50 (Other: IDRCB)
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction, Acute
Keywords: ST-elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+ ICIC + (Experimental): Patients with remote ischemic conditioning and intracoronary ischemic conditioning
  Interventions: Device: Remote ischemic conditioning and intracoronary ischemic conditioning
- RCI - ICIC - (Other): Control group with no remote ischemic conditioning and no intracoronary ischemic conditioning
  Interventions: Device: Patients with no remote ischemic conditioning and no intracoronary ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning and intracoronary ischemic conditioning — RIC: Four cycles of [5 min brachial cuff inflation at 200 mmHg followed by 5 min of cuff deflation] started as soon as possible prior to PCI reperfusion. At least one full cycle (inflation + deflation) has to be completed before PCI reperfusion.
  ICIC: Four cycles of [1 min balloon inflation followed by 1 min balloon deflation] started as soon as possible after reopening of the culprit coronary artery (maximum within 3 minutes after reflow). The balloon will be placed carefully above the culprit lesion so as to minimize potential micro-embolization.
  Arms: RIC+ ICIC +
Device: Patients with no remote ischemic conditioning and no intracoronary ischemic conditioning — Brachial cuff is positioned during 40 minutes but not inflated. No intracoronary balloon inflation.
  Arms: RCI - ICIC -

SUMMARY:
Infarct size is a major determinant of prognosis after AMI. Evidence indicates that the combination of intracoronary ischemic conditioning (ICIC) and remote ischemic conditioning (RIC) can significantly reduce infarct size in STEMI patients. Whether the combination of these two interventions may improve clinical outcome after STEMI remains unknown. The objective of the present study is to determine whether combination of ICIC and RIC can improve STEMI patients clinical outcome at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* All (male and female) patients, aged over 18,
* Presenting within 12 hours of the onset of chest pain,
* For whom the clinical decision was made to treat with percutaneous coronary intervention (PCI),
* ST segment elevation ≥ 0.2 mV in two contiguous ECG leads,
* Written informed consent obtained or oral informed consent certified by a third party.

Non inclusion Criteria:

* Patients with cardiogenic shock,
* Patients with uncontrolled (treated or untreated) hypertension (> 180/110 mmHg),
* Patients with loss of consciousness or confused,
* Patients without health coverage,
* Patient with any legal protection measure,
* Female patients currently pregnant (oral diagnosis) or women of childbearing age who were not using contraception.

Exclusion Criteria:

Patients with main occlusion localized on :

* LAD: distal or ostial segment,
* Non dominant RCA / CX: mid or distal segment,
* Dominant RCA / CX: distal segment,
* Any other arteries apart LAD/CX/RCA; Patients with evidence of coronary collaterals to the risk region (Rentrop score ≥ 2); Patients with an opened (TIMI > 1) culprit coronary artery on initial admission coronary angiography or a failed PCI (final TIMI=0).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Combined incidence of [all-cause mortality; worsening of heart failure during initial hospitalization or re-hospitalization for heart failure at 6 months after MI, large infarct defined as CK peak at 6 hours > 4500 UI/L] | 6 months

SECONDARY OUTCOMES:
Cardiovascular death at 6 months. | 6 months
Worsening of heart failure | 6 months
  Worsening of heart failure during initial hospitalization or re-hospitalization for heart failure at 6 months.
Time to first event [all-cause mortality; worsening of heart failure during initial hospitalization or re-hospitalization for heart failure] | 6 months
Major Adverse Cardiac Events (MACE) | 6 months
  MACE at 6 months: [all-cause mortality; worsening of heart failure during initial hospitalization or re-hospitalization for heart failure; malignant ventricular arrhythmias; recurrent infarction; unstable angina; unplanned revascularization; stroke].
Renal failure | 6 months
  Renal failure (+25% increase in serum creatinine at 6 months versus baseline).
Peak of creatine kinase | 4-6 hours post-PCI
creatine kinase | 5 days
Measure hsCRP | 5 days
Rate of CRP | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rioufol, Pr, Principal Investigator — Hôpital Louis Pradel 28 avenue Doyen Lépine, BP Lyon-Montchat, 69394LYON cedex 03
Locations (4):
- Belgium (3):
  - Algemeen Ziekenhuis Sint Jan, Bruges
  - CHU de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
- Hopital Louis Pradel, Bron, France